CLINICAL TRIAL: NCT06270654
Title: Management of Perioperative Pain Using Erector Spinae Plane Block in Open Microscopic Lumbar Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023322-12280
Record Dates: First submitted 2023-08-28; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Lumbar Spine Disease
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Pre incision of 0.375% ropivacaine 10ml local infiltration will be given.
  Interventions: Procedure: Skin infiltration LA
- Ropivacaine group (Experimental): Bilateral erector spinae plane block (0.375% 20ml ropivacaine on each side + adrenaline 1:200,000) pre incision.
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — After consent was obtained, patients will be randomised into control group and an intervention group. For patients randomized into the interventional group, bilateral erector spinae plane block will be performed under general anaesthesia in prone position before the operation. An experienced anaesthetist performs this under ultrasound guidance (using curvilinear probe) in a sterile method.
  After identifying L3 transverse process, 21G Stimuplex needle will be inserted via in-plane method. Once needle placement is confirmed and aspiration is negative, 20ml of ropivacaine 0.375% with adrenaline 1:200,000 dilution will be given on each side.
  Arms: Ropivacaine group
Procedure: Skin infiltration LA — Pre incision of 0.375% ropivacaine 10ml local infiltration will be given to control group
  Arms: Control group

SUMMARY:
The aim of this study is to compare patients receiving bilateral erector spinae block with ropivacaine vs control group in terms of pain score, total opioid consumption, hemodynamic changes intraoperatively, length of hospitalisation , time to ambulation post surgery and quality of recovery.

DETAILED DESCRIPTION:
Most open spine surgery exacts a high degree of postsurgical pain due to the incision and muscle dissection of the vertebra. The postoperative pain control and early mobilization improve the quality of the surgical care. Inadequate pain relief might result in perioperative morbidity, resulting in prolonged hospital stays.

Erector spinae plane block (ESPB) is an interfascial plane block where local anaesthetic is injected in a plane preferably below the erector spinae muscle. It can provide thoracic, abdominal, and even some lower extremity analgesia. It was also theorised that erector spinae plane block can reduce opioid use and provide analgesia for lumbar surgery. The financial cost that is saved by reducing the length of hospital stay, perioperative morbidity will warrant the use of erector spinae plane block in patients undergoing lumbar spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Patients with Glasgow Coma Scale of 15.
* American Society of Anaesthesiologists (ASA) Physical Status Classification I - II patients
* Scheduled for elective, open microscopic lumbar surgery (less than 3 levels) under general anesthesia.

Exclusion Criteria:

* Cognitive impairment
* Patient refusal
* Weight<50kg, >120kg
* Allergy to local anesthesia
* Alcohol/ drug abuse
* Renal failure or liver failure
* Coagulopathy/thrombocytopenia
* Chronic pain with chronic opioid usage
* Ischemic heart disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain score at recovery, 30mins, 1, 2, 4, 8,12, 24 hours post-surgery | 24 hours
  Measure by numerical rating scale (minimum 1-least pain, maximum 10-most painful)
Total opioid consumption intraoperative | 48 hours
  Measure by total dose consumed (in milligram)
Total opioid consumption post-operative | up to 72 hours
  Measure by total dose consumed (in milligram)
Timing of first rescue dose of iv morphine | up to 24 hours
  Post operation till time requiring first dose of iv morphine

SECONDARY OUTCOMES:
The quality of recovery score (QoR)-15 questionnaire at 24 hours post-operation | 24 hours
  Measure by the quality of recovery score (QoR)-15 questionnaire (minimum of 0,maximum of 150,higher score means a better outcome)
Hemodynamic changes intraoperative | Intraoperative period
  Blood pressure(measure in mm hg)
Hemodynamic changes intraoperative | Intraoperative period
  heart rate (heart rate measure via heart beats per minute/ECG)
Length of hospital stays | up to 1 week
  Days of stay in hospital
Time to ambulation after surgery | up to 1 week
  Time from operation till ambulation

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siddiqui N, Krishnan S, Dua A, Cascella M. Erector Spinae Plane Block. 2025 May 3. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK545305/ PMID 31424889
- [Background] Donnally III CJ, Hanna A, Varacallo MA. Lumbar Degenerative Disk Disease. 2023 Aug 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK448134/ PMID 28846354
- [Background] Kim HS, Wu PH, Jang IT. Lumbar Degenerative Disease Part 1: Anatomy and Pathophysiology of Intervertebral Discogenic Pain and Radiofrequency Ablation of Basivertebral and Sinuvertebral Nerve Treatment for Chronic Discogenic Back Pain: A Prospective Case Series and Review of Literature. Int J Mol Sci. 2020 Feb 21;21(4):1483. doi: 10.3390/ijms21041483. PMID 32098249
- [Background] Grotle M, Smastuen MC, Fjeld O, Grovle L, Helgeland J, Storheim K, Solberg TK, Zwart JA. Lumbar spine surgery across 15 years: trends, complications and reoperations in a longitudinal observational study from Norway. BMJ Open. 2019 Aug 1;9(8):e028743. doi: 10.1136/bmjopen-2018-028743. PMID 31375617
- [Background] Bajwa SJ, Haldar R. Pain management following spinal surgeries: An appraisal of the available options. J Craniovertebr Junction Spine. 2015 Jul-Sep;6(3):105-10. doi: 10.4103/0974-8237.161589. PMID 26288544
- [Background] Tan M, Law LS, Gan TJ. Optimizing pain management to facilitate Enhanced Recovery After Surgery pathways. Can J Anaesth. 2015 Feb;62(2):203-18. doi: 10.1007/s12630-014-0275-x. Epub 2014 Dec 10. PMID 25501696
- [Background] Gan TJ. Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res. 2017 Sep 25;10:2287-2298. doi: 10.2147/JPR.S144066. eCollection 2017. PMID 29026331
- [Background] Jain K, Jaiswal V, Puri A. Erector spinae plane block: Relatively new block on horizon with a wide spectrum of application - A case series. Indian J Anaesth. 2018 Oct;62(10):809-813. doi: 10.4103/ija.IJA_263_18. PMID 30443066
- [Background] Kot P, Rodriguez P, Granell M, Cano B, Rovira L, Morales J, Broseta A, Andres J. The erector spinae plane block: a narrative review. Korean J Anesthesiol. 2019 Jun;72(3):209-220. doi: 10.4097/kja.d.19.00012. Epub 2019 Mar 19. PMID 30886130
- [Background] Canitez A, Kozanhan B, Aksoy N, Yildiz M, Tutar MS. Effect of erector spinae plane block on the postoperative quality of recovery after laparoscopic cholecystectomy: a prospective double-blind study. Br J Anaesth. 2021 Oct;127(4):629-635. doi: 10.1016/j.bja.2021.06.030. Epub 2021 Jul 31. PMID 34340839
- [Background] Vaughan BN, Bartone CL, McCarthy CM, Answini GA, Hurford WE. Ultrasound-Guided Continuous Bilateral Erector Spinae Plane Blocks Are Associated with Reduced Opioid Consumption and Length of Stay for Open Cardiac Surgery: A Retrospective Cohort Study. J Clin Med. 2021 Oct 28;10(21):5022. doi: 10.3390/jcm10215022. PMID 34768541
- [Background] Lin H, Guan J, Luo S, Chen S, Jiang J. Bilateral Erector Spinae Plane Block for Quality of Recovery Following Posterior Lumbar Interbody Fusion: A Randomized Controlled Trial. Pain Ther. 2022 Sep;11(3):861-871. doi: 10.1007/s40122-022-00395-9. Epub 2022 May 23. PMID 35604613
- [Background] Jin Y, Zhao S, Cai J, Blessing M, Zhao X, Tan H, Li J. Erector Spinae Plane Block for Perioperative Pain Control and Short-term Outcomes in Lumbar Laminoplasty: A Randomized Clinical Trial. J Pain Res. 2021 Sep 3;14:2717-2727. doi: 10.2147/JPR.S321514. eCollection 2021. PMID 34512011
- [Background] Zhang TJ, Zhang JJ, Qu ZY, Zhang HY, Qiu Y, Hua Z. Bilateral Erector Spinae Plane Blocks for Open Posterior Lumbar Surgery. J Pain Res. 2020 Apr 5;13:709-717. doi: 10.2147/JPR.S248171. eCollection 2020. PMID 32308470
- [Background] Bhardwaj N. Enhanced recovery after surgery. J Anaesthesiol Clin Pharmacol. 2019 Apr;35(Suppl 1):S3-S4. doi: 10.4103/joacp.JOACP_57_19. No abstract available. PMID 31142952
- [Background] Kaye AD, Urman RD, Rappaport Y, Siddaiah H, Cornett EM, Belani K, Salinas OJ, Fox CJ. Multimodal analgesia as an essential part of enhanced recovery protocols in the ambulatory settings. J Anaesthesiol Clin Pharmacol. 2019 Apr;35(Suppl 1):S40-S45. doi: 10.4103/joacp.JOACP_51_18. PMID 31142958
- [Background] Echeverria-Villalobos M, Stoicea N, Todeschini AB, Fiorda-Diaz J, Uribe AA, Weaver T, Bergese SD. Enhanced Recovery After Surgery (ERAS): A Perspective Review of Postoperative Pain Management Under ERAS Pathways and Its Role on Opioid Crisis in the United States. Clin J Pain. 2020 Mar;36(3):219-226. doi: 10.1097/AJP.0000000000000792. PMID 31868759
- [Background] Neuman MD, Bateman BT, Wunsch H. Inappropriate opioid prescription after surgery. Lancet. 2019 Apr 13;393(10180):1547-1557. doi: 10.1016/S0140-6736(19)30428-3. PMID 30983590
- [Background] Avis G, Gricourt Y, Vialatte PB, Meunier V, Perin M, Simon N, Claret PG, El Fertit H, Lefrant JY, Bertrand M, Cuvillon P. Analgesic efficacy of erector spinae plane blocks for lumbar spine surgery: a randomized double-blind controlled clinical trial. Reg Anesth Pain Med. 2022 Jul 21:rapm-2022-103737. doi: 10.1136/rapm-2022-103737. Online ahead of print. PMID 35863786